CLINICAL TRIAL: NCT06210919
Title: A Phase 1, Single-Center, Single-Arm, Open-Label Study to Evaluate the Safety, Tolerability and Efficacy of Single Dose of TRTP-101 in Adults With Atrophic Scars
Brief Title: Safety and Tolerability of Autologous Adipose-derived Mesenchymal Stem Cells Therapy in Adults With Atrophic Scars
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CellinCells (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIC101-01
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Atrophic Scar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRTP-101 (Experimental): Micro-Block (MiB) manufactured from autologous Adipose-derived Mesenchymal Stem Cells
  Interventions: Biological: TRTP-101

INTERVENTIONS:
Biological: TRTP-101 — Intradermal injection of the each of four sites

SUMMARY:
The purpose of this clinical trial was to evaluate the safety and tolerability for 12 weeks after one dose of TRTP-101 in adults with atrophic scars.

DETAILED DESCRIPTION:
A phase 1 clinical trial to evaluate dose-limiting toxicity by administering a singe dose of TRTP-101 to each of the four sites of atrophic scar.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female aged greater than 19 years
2. Four or more atrophic scars in the joints, genitals, perineum, and face except for the lips, eyes and nose

Exclusion Criteria:

1. History of cell therapy
2. Treatment of Dermal resurfacing, Chemical/Mechanical Peel and Skin Photorejuvenation
3. Treatment of Hyaluronic acid/collagen skin filler, non-permanent soft tissue filler and fat grafting
4. Positive for virus infection
5. Use of Anticoagulant therapy or NSAIDs
6. Thrombocytopenia or other coagulation disorder
7. History of keloid scars
8. Infectious disease or other dermatitis in the area of the atrophic scar
9. Use of Immunosuppressant, immunomodulating drug, anticancer drug or radiation therapy
10. Use of systemic steroid medication
11. History of hypersensitivity or severe allergic reactions (e.g., anaphylaxis, Guillain-Barre syndrome, etc.)
12. Use of retinoid medications

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicity | within 4 weeks
  Dose Limiting Toxicity is defined as Grade ≥ 3 adverse drug reaction according to CTCAE criteria for 4 weeks after administration of TRTP-101

SECONDARY OUTCOMES:
Mean percent change in atrophic scar volume | 1, 4, 8 and 12 weeks
  The depressed volume of atropic scar is measured at baseline and post-treatment visits

CONTACTS AND LOCATIONS:
Overall Officials: Jonghee Lee, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwon HH, Yang SH, Lee J, Park BC, Park KY, Jung JY, Bae Y, Park GH. Combination Treatment with Human Adipose Tissue Stem Cell-derived Exosomes and Fractional CO2 Laser for Acne Scars: A 12-week Prospective, Double-blind, Randomized, Split-face Study. Acta Derm Venereol. 2020 Nov 4;100(18):adv00310. doi: 10.2340/00015555-3666. PMID 33073298
- [Background] Cho YB, Lee WY, Park KJ, Kim M, Yoo HW, Yu CS. Autologous adipose tissue-derived stem cells for the treatment of Crohn's fistula: a phase I clinical study. Cell Transplant. 2013;22(2):279-85. doi: 10.3727/096368912X656045. Epub 2012 Sep 21. PMID 23006344
- [Background] Salloum RH, Rubin JP, Marra KG. The role of steroids in mesenchymal stem cell differentiation: molecular and clinical perspectives. Horm Mol Biol Clin Investig. 2013 Aug;14(1):3-14. doi: 10.1515/hmbci-2013-0016. PMID 25436715